CLINICAL TRIAL: NCT03302611
Title: A Randomized Controlled Trial of Surf and Hike Therapy for Active-duty Service Members With Major Depressive Disorder
Brief Title: Trial of Surf and Hike Therapy for Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Collaborators: Naval Health Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kristen Walter, Clinical Research Psychologist, United States Naval Medical Center, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMCSD.2017.0007
Record Dates: First submitted 2017-10-02; First posted 2017-10-05 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Major Depressive Disorder
Keywords: major depressive disorder; military; surf therapy; hike therapy; randomized controlled trial
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Consenting active duty service members with major depressive disorder will be randomized to receive 6 weeks of either surf or hike therapy. Participants will be allowed to receive the other intervention (i.e., the condition that they were not originally randomized to) if interested after the initial intervention period.
Who Masked: Outcomes Assessor
Masking Description: The assessor will be blinded to participants' intervention condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surf Therapy (Experimental): Participants receive a physical activity-based intervention, which in this arm is surf therapy. Each service member is paired with a surf instructor who typically works with them each week for the length of the program.
  Interventions: Behavioral: Physical Activity-based Interventions
- Hike Therapy (Active Comparator): Participants receive a physical activity-based intervention, which in this arm is hike therapy. During hike therapy, service members may hike together or at a self-selected pace.
  Interventions: Behavioral: Physical Activity-based Interventions

INTERVENTIONS:
Behavioral: Physical Activity-based Interventions — Participants will be randomized to one of two physical activity-based interventions, surf or hike therapy.

SUMMARY:
This study uses a randomized controlled trial design to compare the psychological effects of surf therapy to hike therapy in active duty service members who have been diagnosed with major depressive disorder.

DETAILED DESCRIPTION:
This prospective, longitudinal randomized controlled trial will enroll up to 86 active duty service members with major depressive disorder who are seeking surf or hike therapy as part of their standard medical care. Participants will be randomly assigned to receive 6 weeks of either surf or hike therapy. Assessor-administered and self-report measures will be completed at pre- and post-program, as well as three months following program completion. Participants also will complete brief, self-report assessments before and after each program activity session.

ELIGIBILITY:
Inclusion Criteria:

* Be a military service member seeking surf or hike therapy as part of the Wounded, Ill, and Injured Wellness program at Naval Medical Center San Diego;
* Have medical clearance to participate in these programs;
* Have a current diagnosis of Major Depressive Disorder based on DSM-5 criteria.

Exclusion Criteria:

* Service members who are currently receiving surf or hike therapy (i.e., have already started attending program sessions);
* Service members who are currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | 5 months
  The MADRS is a widely used, semi-structured, clinical-interview assessment of depression symptom severity that is intended to be sensitive to change following an intervention.

SECONDARY OUTCOMES:
PTSD Checklist (PCL-5) | 5 months
  The PCL-5 is a self-report instrument assessing PTSD symptom severity.
Generalized Anxiety Disorder (GAD-7) | 5 months
  The GAD-7 is a self-report instrument that assesses the presence and severity of generalized anxiety disorder.
Short Form Health Survey - 36 Item, Version 2 (SF-36) | 5 months
  The SF-36 is a widely used questionnaire that assesses functioning physical and mental health based on eight summary measures.
Positive and Negative Affect scales (PANAS) | 5 months
  PANAS is a self-report instrument that measures the extent of 20 feelings and emotions experienced within the past few hours.
Insomnia Severity Index (ISI) | 5 months
  The ISI is a 7-item self-report measure that assesses the nature, severity, and impact of insomnia.
Patient Health Questionnaire (PHQ-9) | 5 months
  The PHQ-9 is a self-report instrument that assesses the presence and severity

OTHER OUTCOMES:
Pain Rating Scale (PRS) | 5 months
  The PRS is a self-report measure that assesses current level of pain. It consists of one item rated on an 11-point scale from 0 (no pain) to 10 (worst possible pain).

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia J. Thomsen, Ph.D., Principal Investigator — Naval Health Research Center
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walter KH, Otis NP, Glassman LH, Ray TN, Michalewicz-Kragh B, Kobayashi Elliott KT, Thomsen CJ. Comparison of surf and hike therapy for active duty service members with major depressive disorder: Study protocol for a randomized controlled trial of novel interventions in a naturalistic setting. Contemp Clin Trials Commun. 2019 Aug 21;16:100435. doi: 10.1016/j.conctc.2019.100435. eCollection 2019 Dec. PMID 31485546
- [Result] Walter KH, Otis NP, Ray TN, Glassman LH, Beltran JL, Kobayashi Elliott KT, Michalewicz-Kragh B. A randomized controlled trial of surf and hike therapy for U.S. active duty service members with major depressive disorder. BMC Psychiatry. 2023 Feb 17;23(1):109. doi: 10.1186/s12888-022-04452-7. PMID 36805672
- [Result] Otis NP, Walter KH, Glassman LH, Ray TN, Kobayashi Elliott KT, Michalewicz-Kragh B. Comorbidity of depression and posttraumatic stress disorder: Outcomes from a randomized controlled trial of surf and hike therapies among service members. Psychol Trauma. 2024 Dec;16(Suppl 3):S688-S697. doi: 10.1037/tra0001673. Epub 2024 Jul 8. PMID 38976384
- [Result] Glassman LH, Otis NP, Kobayashi Elliott KT, Michalewicz-Kragh B, Walter KH. Gender Differences in Psychological Outcomes Following Surf versus Hike Therapy among U.S. Service Members. Int J Environ Res Public Health. 2024 Feb 19;21(2):241. doi: 10.3390/ijerph21020241. PMID 38397730
- [Result] Walter KH, Otis NP, Miggantz EL, Ray TN, Glassman LH, Beltran JL, Kobayashi Elliott KT, Michalewicz-Kragh B. Psychological and functional outcomes following a randomized controlled trial of surf and hike therapy for U.S. service members. Front Psychol. 2023 Jun 8;14:1185774. doi: 10.3389/fpsyg.2023.1185774. eCollection 2023. PMID 37359884
- See also: Link to outcomes manuscript — https://doi.org/10.1186/s12888-022-04452-7